CLINICAL TRIAL: NCT01899378
Title: Safety and Efficacy of Probiotics in Bangladeshi Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Julie Parsonnet, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SPO109949
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- daily probiotic (Experimental): 10^8 CFU Lactobacillus reuteri DSM 17938 and 10^9 Bifidobacterium longum infantis daily for one month
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938; Dietary Supplement: Bifidobacterium longum infantis
- weekly probiotic (Experimental): 10^8 CFU Lactobacillus reuteri DSM 17938 and 10^9 Bifidobacterium longum infantis weekly for one month
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938; Dietary Supplement: Bifidobacterium longum infantis
- bi-weekly probiotic (Experimental): 10^8 CFU Lactobacillus reuteri DSM 17938 and 10^9 Bifidobacterium longum infantis bi-weekly for one month
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938; Dietary Supplement: Bifidobacterium longum infantis
- control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — 10^8 CFU
  Other Names: BioGaia Protectis Baby
  Arms: bi-weekly probiotic; daily probiotic; weekly probiotic
Dietary Supplement: Bifidobacterium longum infantis — 10^9 CFU
  Other Names: Align
  Arms: bi-weekly probiotic; daily probiotic; weekly probiotic

SUMMARY:
Here the investigators propose to preliminarily investigate the safety and effects of probiotics in infants in Bangladesh through a pilot randomized clinical trial. The investigators hypothesize that two probiotics are safe for infants in Bangladesh and may have an effect on biomarkers of gut health and immunity. The specific aims of this pilot are: i) to confirm the safety of administering probiotic strains to infants in low-income countries, ii) to determine the effects of dosing frequency on colonization and persistence of probiotics in the GI tract, iii) to measure markers of intestinal and immune function and microbiota structure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants.
* Infants 1 -3 months of age at the beginning of the study.
* Parents/guardians of each subject are able to understand study procedures and agree to participate in the study by giving consent.
* Parents and child are planning to remain in Dhaka for the next four months.

Exclusion Criteria:

* Infants with known birth defects.
* Infants who have been hospitalized.
* Infants who have an acute infection or illness at the time of enrolment.
* Infants who are currently taking antibiotics
* Infants <1 month of age or >3 months of age.
* Infants three standard deviations below mean on anthropometric measures (will be referred for medical care).
* Infants who are already receiving a probiotic product or treatment.
* A diagnosis or suspicion of immunodeficiency disorder.
* A diagnosis or suspicion of bleeding disorder that would contraindicate venipuncture.
* Family residence outside of Dhaka or families expecting to move outside of Dhaka in the next 4 months.

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Presence of probiotic in the stool | weeks 0-12
  presence of absence of each probiotic in the stool
Adverse events | duration of study - through study completion
  Any adverse or allergic reactions after probiotic administration, hospitalizations, GI and respiratory symptoms

SECONDARY OUTCOMES:
quantity of probiotic in the stool | weeks 0-12
  amount of each probiotic present in the stool
composition of microbiota | weeks 0-12
  microbial community composition
clinical effects | daily for 7 days after first probiotic administration, then weeks 2-12
  fever, diarrhea, wheezing, rash, stool frequency, feeding frequency
gut function | months 0, 1, 2, 3
  lactulose/mannitol ratio
gut inflammation | months 0,1,2,3
  fecal neopterin, alpha-1 antitrypsin, and myeloperoxidase - correlated with future growth
gut inflammation/translocation | months 0, 1, 2, 3
  IL22, CD-14, total IgG and c-reactive protein
growth | month 0, 1, 2, 3
  weight, length, head circumference
breastfeeding rates | month 0, 1, 2, 3

CONTACTS AND LOCATIONS:
Overall Officials: Yana Emmy E Hoy-Schulz, PhD, Study Director — Stanford University; Julie Parsonnet, MD, Principal Investigator — Stanford University; Stephen Luby, MD, Principal Investigator — Stanford University; Leanne Unicomb, PhD, Principal Investigator — International Center for Diarrheal Disease Research, Bangladesh; Kaniz Jannat, MBBS, Study Director — International Center for Diarrheal Disease Research, Bangladesh
Locations (1):
- International Center for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Roberts TJ, Hoy-Schulz YE, Jannat K, Parsonnet J. Evidence of inflated exclusive breastfeeding estimates from a clinical trial in Bangladesh. Int Breastfeed J. 2018 Aug 22;13:39. doi: 10.1186/s13006-018-0179-4. eCollection 2018. PMID 30159001
- [Derived] Hoy-Schulz YE, Jannat K, Roberts T, Zaidi SH, Unicomb L, Luby S, Parsonnet J. Safety and acceptability of Lactobacillus reuteri DSM 17938 and Bifidobacterium longum subspecies infantis 35624 in Bangladeshi infants: a phase I randomized clinical trial. BMC Complement Altern Med. 2016 Feb 2;16:44. doi: 10.1186/s12906-016-1016-1. PMID 26832746